CLINICAL TRIAL: NCT05862090
Title: An Open Label, Multiple Dose, Crossover Clinical Trial to Evaluate the Drug-drug Interaction and Safety of RLD2301 and RLD2007 After Oral Administration in Healthy Volunteers
Brief Title: A Study to Evaluate the Drug-drug Interaction and Safety of RLD2301 and RLD2007 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ENSEMBLE-101
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (First RLD2301, then RLD2301+RLD2007) (Experimental): Period1 : RLD2301 Period2 : RLD2301 + RLD2007
  Interventions: Drug: RLD2301; Drug: RLD2007
- Arm 2 (First RLD2007, then RLD2301+RLD2007) (Experimental): Period1 : RLD2007 Period2 : RLD2301 + RLD2007
  Interventions: Drug: RLD2301; Drug: RLD2007

INTERVENTIONS:
Drug: RLD2301 — Take it once a day per period.
Drug: RLD2007 — Take it once a day per period.

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction and safety of RLD2301 and RLD2007 after oral administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~54 years in healthy volunteers
* 18.5 kg/m^2 ≤ BMI < 30 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <90 mmHg
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
AUCtau | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
Css,max | 0~24 hours after final dose administration
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
Css,min | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
Css,av | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
Tss,max | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
t1/2 | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
CLss/F | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
Vdss/F | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
Fluctuation[(Css,max-Css,min)/Css,av] | 0~24 hours after final dose administration
  Pharmacokinetic evaluation
Swing[(Css,max-Css,min)/Css,min] | 0~24 hours after final dose administration
  Pharmacokinetic evaluation

OTHER OUTCOMES:
Change of Blood Pressure(SBP/DBP) from baseline | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
Change of pulse rate from baseline | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
Change of blood glucose from baseline | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
AUECtau of Blood Pressure(SBP/DBP) | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
AUECtau of pulse rate | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
AUECtau of blood glucose | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
Emax of Blood Pressure(SBP/DBP) | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
Emax of pulse rate | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation
Emax of blood glucose | Predose at Day1 and 0~24 hours after final dose administration of each period
  Pharmacodynamic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, MD, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk University Hospital, Jeonju, Jeollabuk-do, South Korea